CLINICAL TRIAL: NCT07336836
Title: Characterization of the Effects of Oral NAD+ in a Wellness Cohort
Brief Title: Renewal-NAD+: A Study of Oral NAD+ and Its Multi-omic Impact in a Healthy Cohort
Acronym: Renewal-NAD+
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: BioNADrx Holdings, Inc. Bryleos (Industry)
Collaborators: ISB Analytica, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1320748
Record Dates: First submitted 2025-12-19; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Health Adult Subjects; Healthy Participants
Keywords: NAD+, dietary supplement

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study was double blinded, all investigators, study personnel, molecular facilities and participants were naive to treatment identity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): LNAD+ (50%)/PEG (50%) treatment total 500 mg
  Interventions: Dietary Supplement: LathMized TM NAD+ (LNAD+)
- Control arm (Placebo Comparator): PEG 500 mg
  Interventions: Other: Control (placebo)

INTERVENTIONS:
Dietary Supplement: LathMized TM NAD+ (LNAD+) — NAD+ 500 mg
  Arms: Treatment arm
Other: Control (placebo) — PEG (100% of mass)
  Arms: Control arm

SUMMARY:
The goal of this 5 day interventional study was to investigate the effects on multiple biological molecules (multi-omics) of Bryleos's commercially available oral LathMized™ Nicotinamide adenine dinucleotide (LNAD+) supplement in healthy adults aged 45-75 years. The main question to be answered was whether LNAD+ supplementation is associated with change in biological markers relevant to subjects' health. Also, the study determined whether this oral NAD+ formulation raised NAD+ levels including inside blood cells, after the 5 day treatment period, measured on post-treatment Day 1 (Day 6). Thus, the study compared NAD+ levels and impact on biological markers in the LNAD+ arm versus control placebo arm. Safety in this population was assessed using clinical laboratory tests, daily self-reporting of symptoms, and data from a wearable device.

DETAILED DESCRIPTION:
The RENEWAL-NAD+ study was designed as a single-center (distributed) Phase 0/1 double-blind, randomized, placebo-controlled clinical trial to evaluate the safety, tolerability, and pharmacodynamic effects of five days of oral LNAD+ (LathMized™ NAD+) in healthy aging adults aged 45 to 75 years (inclusive).

The Renewal-NAD+ study was motivated by the dearth of evidence on oral NAD+ bioavailability and current limited understanding of the mechanisms of action and multi-omic footprint of NAD metabolism interventions from a systems biology standpoint. The present first-in-humans study was designed as a key translational step in establishing the safety, tolerability, and biological effects of LNAD+ in human subjects. The study aimed to demonstrate that theoretical advantages and documented preclinical benefits of enhanced NAD+ delivery translate to meaningful biological changes in healthy aging humans. It also provides meaningful data on the broader biological implications of NAD repletion that could translate into improvements in a multitude of therapeutic areas.

The novel formulation of NAD+ (LNAD+) had been commercially available prior to study initiation and was developed as a systematic formulation approach to the multifaceted barriers that have prevented effective oral NAD+ delivery. The proprietary LathMize™ Technology stabilizes and protects NAD+ before and during GI transit while facilitating absorption through multiple complementary mechanisms including optimizing particle size distribution to enable uptake through multiple pathways.

The study examined the effects of oral LNAD+ supplementation on intracellular and circulating NAD+ levels, as well as on levels of peripheral blood biomarkers, vitals, patient-reported outcomes, activity and sleep measures obtained via a wearable fitness device, and frequency of adverse events in a cohort of healthy adults The study aimed to enroll 60 adults in overall good health to obtain four longitudinal blood draws (two baseline and two on-treatment, respectively) and examined changes in circulating and intracellular NAD+, clinical laboratory tests, and plasma proteome and metabolome composition, in the LNAD+ arm relative to placebo.

The study was designed as a one-center but distributed trial that relied on the combination of ISB BioAnalytica's proprietary Electronic Data Capture (EDC) platform, at-home supplementation by the study participants, and mobile phlebotomy visits for venipuncture and vitals collection.

The study protocol was divided into 3 sequential phases:

Phase I: Screening/Eligibility. Phase II: Treatment Allocation and Wash-out. Phase III: Masked Treatment.

The study enrolled adults age 45-75 without pre-specified targeted health conditions with the following objectives:

1. The primary objective was to demonstrate the bioavailability of orally administered LNAD+ through measurement of both intracellular and extracellular NAD+ concentrations. This dual assessment approach recognizes that systemic NAD+ levels may not accurately reflect cellular delivery. Specifically, the selection of intracellular measurements in peripheral blood mononuclear cells provides direct evidence of cellular NAD+ augmentation rather than systemic exposure. The temporal assessment strategy captures both short-term responses and steady-state achievement, enabling characterization of pharmacokinetic and pharmacodynamic profiles.
2. Complementing this primary objective, the secondary objectives encompass comprehensive short-term safety evaluation and mechanistic characterization of LNAD+ through targeted biomarker assessment. The safety evaluation included analysis of adverse events, daily reports of physiological symptoms by body system, and detailed laboratory assessment of hepatic, renal, and hematological parameters, recognizing that metabolic interventions may have subtle systemic effects, as well as data obtained from a wearable device. The pharmacodynamic biomarker panel spanned multiple biological systems identified as responsive to NAD+ in preclinical studies, including inflammatory markers, metabolic parameters (lipid profiles, glucose metabolism), kidney and liver function markers, reactive oxidative species, and potential safety-related biomarkers .
3. The exploratory objective was to characterize the systems-level effects of NAD+ augmentation in humans through comprehensive multi-omic profiling of peripheral blood samples. High-throughput plasma metabolomics characterized the metabolic fate of administered NAD+ and identified downstream metabolic reprogramming. Proteomic profiling using high-throughput targeted discovery proteomics evaluated changes in circulating proteins relevant to inflammation, metabolism, and cellular stress responses. This unbiased discovery approach was designed to also identify novel candidate biomarkers of NAD+ response and potentially identify subpopulations most likely to benefit from intervention.

ELIGIBILITY:
Inclusion Criteria: English-speaking adults in the age range between 45 and 75 years in overall self-reported good health (excluding common conditions such as hypertension, and hyperlipidemia);

* Participants able to consent for themselves;
* Able to commit to the study protocol, including a 7-day washout of potentially confounding substances via restriction of supplement intake;
* Tolerance for repeated venous blood draws, supplement administration, and assessment schedule, tolerance for wrist-worn wearable devices well (i.e., consistent use during the day as well as at night for the duration of the study).

Exclusion Criteria:

* Body Mass Index (BMI) > 35 kg/m2;
* Current chronic or acute infectious diseases (e.g., hepatitis, influenza, HIV, Lyme; COVID-19 within the past two months);
* Recent SARS-CoV-2 vaccine administration (within two weeks);
* Current use of NAD+ supplements and precursors;
* Use of systemic anti-inflammatory medications (excluding NSAIDs and acetaminophen), immunosuppressants;
* Current cancer or hematologic conditions and/or cancer treatment (radiation, chemotherapy);
* Type I juvenile or Type 2 diabetes mellitus;
* Autoimmune disorders (multiple sclerosis, lupus, rheumatoid arthritis, psoriasis);
* Inflammatory bowel disease (ulcerative colitis, Crohn's disease);
* Current pregnancy;
* Current substance abuse, including alcohol, but excluding nicotine and prescription medications (e.g., physician-prescribed stimulants, opiates);
* Members of the same household.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2022-06-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics-NAD+ concentrations | From enrollment through seven day washout, 2 baseline measurements); treatment 5 days, measured on day 3 and one day post day 5 treatment (Day 6)]
  All primary endpoint NAD+ measurements were performed by a CLIA-certified laboratory (Augusta, GA, USA). The proprietary validated enzymatic assay quantifies total NAD (NAD+ plus NADH) in both intracellular (icNAD) and circulating (cirNAD) compartments. The assay specifically quantifies total NAD, reflecting technical considerations and the current state of clinical validation for NAD+/NADH ratio measurements. For most clinical applications, including assessment of supplementation efficacy, total NAD levels can be considered the primary actionable biomarker.

SECONDARY OUTCOMES:
Pharmacodynamic Endpoints: Metabolic Fate | From enrollment through seven day washout, (2 baseline measurements); treatment 5 days, measured on day 3 and one day post day 5 treatment (Day 6)
  Metabolic fate: plasma abundance of six NAD+ metabolites was assayed via Metabolon's Global Discovery Platform, including nicotinamide (NAM), methylated NAM (MeNAM), 2PY, nicotinate, trigonelline, and quinolinate.
  •
Pharmacodynamic Endpoints:Liver Function | From enrollment through seven day washout, (2 baseline measurements); treatment 5 days, measured on day 3 and none day post day 5 treatment (Day6)]
  Serum alanine transaminase, aspartate transaminase, alkaline phosphatase, and total bilirubin
Pharmacodynamic Endpoints: Oxidative Stress | From enrollment through seven day washout, (2 baseline measurements); treatment 5 days, measured on day 3 and none day post day 5 treatment (Day6)]
  Oxidative stress: gamma glutamyl transferase and cumulative reactive oxygen metabolites (ROM) were used as surrogate endpoints. Cumulative ROM included oxygen O2, superoxide anion O2-, peroxide O2-, hydrogen peroxide H2O2, hydroxyl radical OH, and hydroxyl ion OH-.
Pharmacodynamic Endpoints: Glucose Metabolism | From enrollment through seven day washout, 2 baseline measurements); treatment 5 days, measured on day 3 and one day post day 5 treatment (Day 6)]
  Glucose metabolism: fasting serum glucose.
Pharmacodynamic Endpoints: Lipid Metabolism | From enrollment through seven day washout, (2 baseline measurements); treatment 5 days, measured on day 3 and one day post day 5 treatment (Day 6)
  Lipid metabolism: serum triglycerides, LDL, HDL, and HDL/LDL ratio.
Pharmacodynamic Endpoints: Inflammation | From enrollment through seven day washout, 2 baseline measurements); treatment 5 days, measured on day 3 and one day post day 5 treatment (Day 6)]
  Inflammation: indexed by a combination of pro-inflammatory cytokines TNF, IL-6, and hs-CRP, as well complete blood count differentials.
Pharmacodynamic Endpoint: Kidney Function | From enrollment through seven day washout, (2 baseline measurements); treatment 5 days, measured on day 3 and none day post day 5 treatment (Day6)]
  Kidney Function: serum creatinine, estimated glomerular filtration rate (eGFR) and blood urea nitrogen
Physical Safety Measures: Vitals | From enrollment to end of treatment day 5 (measured post treatment Day 1(Day 6)]
  Vitals: Height and weight, BMI (kg/m3) were measured twice and averaged for each study blood draw / mobile phlebotomist visit. •
  :
Physical Safety Measures: Vitals | Time Frame: From enrollment to end of treatment day 5 (measured post treatment Day 1 [Day6])
  Systolic and diastolic blood pressure (mm/Hg and resting heart rate (bpm) were measured twice and averaged for each study blood draw / mobile phlebotomist visit.
Physical Safety Measures: Adverse Events | From enrollment to end of treatment day 5 (measured post treatment Day 1[Day6]
  Patient-reported adverse event incidence was tabulated at the end of the study
Physical Safety Measures: Physical Symptoms | From enrollment to end of treatment day 5 (Measured post treatment day 5 [Day6])
  Daily self-reported physical symptom data across body and organ system
Physical Safety Measures: subjective measures of well-ing | From enrollment to end of treatment day 5 (Measured post treatment day 5 [Day6])
  Administered self-report questionnaires including a daily version of Depression, Anxiety, and Stress Scale 21 or DASS-21, with appropriate modifications given the design of the study; Clinically Useful Anxiety Outcome Scale-Daily Version or CUXOS-D
Physical Safety Outcome Measures: Wearables Data | From first day of study washout period to end of treatment day 5 (Measured post treatment day 5 [Day6])
  Wearable data were collected using Fitbit Luxe devices. Examined surrogate endpoints included indices of activity (steps) and sleep quality

OTHER OUTCOMES:
Exploratory Biological Molecules (Multi-omics) | From enrollment through seven day washout, 2 baseline measurements); treatment 5 days, measured on day 3 and one day post day 5 treatment (Day 6)]
  Participants' blood samples were comprehensively profiled using two advanced high-throughput molecular assaying platforms aimed at characterizing the impact of LNAD+ on the plasma metabolome and proteome. Plasma metabolome assaying was performed by Metabolon. Plasma proteome was assayed using the Olink Explore platform by the core facility at Institute for Systems Biology (Seattle, WA).

CONTACTS AND LOCATIONS:
Locations (1):
- ISB Bioanalytica, Inc., Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No